CLINICAL TRIAL: NCT05802966
Title: Cognition in Mindfulness: Negativity and Depression
Acronym: CogMiND
Status: Terminated | Type: Observational
Why Stopped: No (financial) means left to continue inclusion to achieve predetermined sample size. Instead of continuation (high probability of unanalyzed data) it was decided to stop inclusion and analyze data, so the scientific community can benefit from it.
Sponsor: Radboud University Medical Center (Other)
Collaborators: Pro Persona Mental Health Care Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: NL68398.091.18
Record Dates: First submitted 2023-03-09; First posted 2023-04-07 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-03

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Mindfulness-Based Cognitive Therapy; Working mechanisms
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mindfulness-Based Cognitive Therapy + Treatment as usual: Patients receive Mindfulness-Based Cognitive Therapy (MBCT) and treatment as usual (TAU). Measurements are administered before, half-way and after MBCT.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy
- Wait-list control (Treatment as usual): Patients in the wait-list controlled group receive treatment us usual (TAU) during their waiting-period. After their waiting period, they receive MBCT in a similar fashion compared to the intervention group. Measurements are administered before, half-way and after their waiting period. In addition, a fourth and fifth measurement will be administered half-way and after MBCT.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy — MBCT will be offered according to the MBCT manual developed for relapse prevention in MDD (Zindel V. Segal, Williams, & Teasdale, 2002). Thus, MBCT will consist of 8-weekly sessions of 2,5 hours, a 6-hour silent day, and daily home practice (± 45min). MBCT will be taught by a certified MBCT teacher meeting the advanced criteria of the Association of Mindfulness Based Teachers in the Netherlands and Flanders (Belgium) which are in concordance with the Good Practice guidelines of the UK Network of Mindfulness-Based Teacher Trainers (Crane et al., 2012).

SUMMARY:
Mindfulness-Based Cognitive Therapy (MBCT) is effective in reducing relapse rates and (residual) symptoms in major depressive disorder (MDD). However, the mechanisms underlying those MBCT-induced effects are far from clear. The goal of this study is to get more insight into the working mechanisms of MBCT. The main question to be answered is whether MBCT-induced reduction in depressive symptoms is mediated and/or moderated by repetitive negative thinking (RNT), or other factors hypothesized to be involved in the working mechanism of MBCT (e.g. mindfulness skills and self-compassion).

DETAILED DESCRIPTION:
Introduction

Depression is highly prevalent and is ranked by the world health organization (WHO) as the number one contributor to disability worldwide. The highly recurrent nature of the disorder contributes greatly to the burden of Major Depressive Disorder (MDD) and with every new depressive episode, outcome prospective worsen. Mindfulness Based Cognitive Therapy (MBCT) is an effective treatment to reduce relapse rates and (residual) symptoms that contribute to recurrence in MDD. However, the mechanisms underlying this MBCT-induced effect are far from clear.

Elucidating these mechanisms will provide insight in the existing individual differences in effectiveness of MBCT. Consequently, this insight will help to improve effectiveness of treatment and even personalize treatment regimes. One likely candidate that could play a major role in the positive effects of MBCT on depressive symptoms, is repetitive negative thinking (RNT). Depressive rumination is the most well-studied form in the context of depression and has been described as the process of thinking perseveratively about one's feelings and problems (such as symptoms of depression) and their possible causes and consequences. It is believed that during MBCT participants develop the ability to become aware of automatic maladaptive cognitive processes such as depressive rumination, and learn to decenter and disengage from them. Because of this core skill to be learned during MBCT patients may be prevented to enter a vicious cycle of ruminative thinking that could otherwise aggravate symptoms of depression or have resulted in a new depressive episode.

Objectives

Our main objectives are (i) to replicate the beneficial effects of MBCT on depressive symptoms and RNT in patients with chronic or recurrent depression (crMDD), and (ii) to investigate whether individual levels of RNT (iia) mediate and/or (iib) moderate the MBCT-induced reduction in depressive symptoms.

To this end self-report questionnaires of depressive symptoms, content-independent RNT and depressive rumination will be administered before, half-way and after MBCT (intervention group) or before, half-way and after a waiting-period (waitlist group).

Secondary objectives

To triangulate research findings an experimental task (breathing focus task) that measures intrusive thoughts during task performance will be administered.

Moreover, research will focus on cognitive control and affective biases therein, because this process is related to RNT. Two major constituents of cognitive control will be measured, i.e. working memory processing and motivational biases of cognitive control (with respectively a working-memory update/ignore emotion task and Pavlovian-to-instrumental transfer task) before and after MBCT/waitlist. This behavioural data will be used to assess whether working memory and motivational biases are indeed (i) related to RNT and MDD, (ii) are changed by MBCT and (iii) whether these changes are related to clinical effects of MBCT.

Additionally, the timing of change will be investigated by administering weekly self-report questionnaires.

Design:

A multicenter, wait-list controlled-trial, with assignment to an intervention group (MBCT + treatment as usual (TAU)) or waitlist-control group (TAU) based on date of intake and start date of MBCT. Thus, assignment is not randomized and the study does not interfere with regular clinical practice (e.g. planning MBCT). If patients have to wait > 7 weeks for the next MBCT, they are invited to participate in the wait-list group while patients that have to wait < 7 weeks will be assigned to the intervention group. Note that although a full MBCT-training training lasts 8 weeks, for feasibility a cut-off of 7 weeks instead of 8 was deliberately chosen because this allows us to assign more patients to the wait-list group. This was done to prevent (as much as possible) an anticipated skewed allocation in favour of the intervention group.

Healthy controls will be invited to one measurement as a benchmark for the innovative cognitive tasks and do not follow MBCT.

Statistical analysis:

A detailed description of the planned analyses can be found within the attached Statistical Analysis Plan.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18
* diagnosis of chronic or recurrent MDD according to DSM-V criteria, both current or remitted
* able to give informed consent and perform experimental tasks

Exclusion Criteria:

* in remission of first (not chronic) episode or having a first (not chronic) current episode
* insufficient comprehension of the Dutch language
* physical, cognitive, or intellectual impairments interfering with participation such as deafness, blindness, or sensorimotor handicaps
* formerly involved in MBCT or MBSR or other 8-week Mindfulness-Based Intervention (MBI)
* meets criteria for bipolar disorder, schizophrenia, schizophreniform disorder, schizoaffective illness or anorexia nervosa
* current psychosis
* high level of suicidality
* drug or alcohol addiction in the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic or recurrent MDD who are referred for MBCT at the RadboudUMC Centre for Mindfulness or at different locations of a local mental health institute (Pro Persona) will be recruited for the current study. Those patients will follow regular medical intake-procedures in accordance to procedures at the respective institutes and are screened for chronic or recurrent depression and other in- and exclusion criteria. Depression will be considered chronic if patients meet the DSM-V criteria of a 'persistent depressive disorder', which is combination of the 'chronic depressive disorder' and 'dysthymic disorder' as defined in the DSM-IV.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | Change from baseline to mid-treatment (4 weeks), to post-treatment (8 weeks)
  Measured with the Inventory of Depressive Symptomatology Self-Report (IDS-SR). The IDS-SR consists of 30 items. Scores range from 0-84. Higher scores indicate a higher severity of depression.
Depressive rumination | Change from baseline to mid-treatment (4 weeks), to post-treatment (8 weeks)
  Measured with the brooding subscale of the Ruminative Response Scale (RRS). The brooding subscale consists of 5 items. Scores range from 5-20. Higher scores indicate a higher level of depressive rumination.
Repetitive negative thinking (RNT) | Change from baseline to mid-treatment (4 weeks), to post-treatment (8 weeks)
  Measured by the Perseverative Thinking Questionnaire (PTQ). The PTQ consists of 15 items. Scores range from 0-60. Higher scores indicate a higher level of repetitive negative thinking.

SECONDARY OUTCOMES:
Intrusive thoughts (state measure) | Change from baseline to mid-treatment (4 weeks), to post-treatment (8 weeks)
  Measured with the breathing focus task (BFT) that measures negative, positive and neutral thoughts during task performance
Mindfulness Skills | Change from baseline to mid-treatment (4 weeks), to post-treatment (8 weeks)
  Measured with the Five Facet Mindfulness Questionnaire - Short Form (FFMQ-SF). This questionnaire is divided into the subscales observing (4 items), and describing, acting with awareness, non-judging and non-reactivity (all 5 items). The facets scores will be calculated by determining the mean of corresponding item scores. Negatively-phrased items will be reversed scored before computing the mean scores of the subscales. Subscale scores range from 1-5, with higher scores indicating 'higher/better' ability of mindfulness on the corresponding domain.
Anxiety Symptoms | Change from baseline to mid-treatment (4 weeks), to post-treatment (8 weeks)
  Measured with the Spielberger State-Trait Anxiety Inventory (STAI). The STAI consists of 20 items. Scores range from 20-80. Higher scores indicate a higher severity of anxiety.
Overall functioning | Change from baseline to mid-treatment (4 weeks), to post-treatment (8 weeks)
  Measured with the Outcome Questionnaire - 45 (OQ-45). The OQ-45 consists of 45 items. Scores range from 0-180. Higher scores indicate higher symptom severity.
Self-compassion | Change from baseline to mid-treatment (4 weeks), to post-treatment (8 weeks)
  Measured with the Self Compassion Scale - Short form (SCS-SF). The scale consists of six subscales each containing 2 items: self-kindness, self-judgment, common humanity, isolation, mindfulness and over-identification. The negatively phrased items will be reversed-scored before calculating subscale and total scores. Each subscale ranges from 2-14. A higher score indicates a higher level (better outcome) of self-kindness, common humanity, mindfulness, self-judgment, isolation, and over-identification. Total scores range from 12 to 84 (summed subscale scores), a higher score indicates a higher level of self-compassion.
Influence of Pavlovian information on goal-directed behaviour | Change from baseline to mid-treatment (4 weeks), to post-treatment (8 weeks)
  Measured with the Pavlovian to Instrumental Transfer (PIT) task
Working memory - emotion-dependent update and ignore capacity of working memory | Change from baseline to mid-treatment (4 weeks), to post-treatment (8 weeks)
  Measured with the Working Memory Update/Ignore Emotion Task (WMUIET)

OTHER OUTCOMES:
Depressive symptoms | Week-to-week change assessed after each MBCT session (up to 8 weeks) or weekly during wait-list (up to 8 weeks)
  Measured with the Quick Inventory of Depressive Symptomatology Self-Report (QIDS-SR). The QIDS-SR consists of 16 items. Scores range from 0-27. Higher scores indicate a higher severity of depression.
Non-judging mindfulness skill | Week-to-week change assessed after each MBCT session (up to 8 weeks) or weekly during wait-list (up to 8 weeks)
  Measured with the non-judging subscale of the FFMQ. This subscale consists of 8 items. Negatively-phrased items will be reversed-scored before calculation of either (i) a sumscore of all items (range 8-40), or the mean of the subscale (range 1-5). A higher score indicates a better/higher capability of the non-judging domain of mindfulness.
Depressive rumination | Week-to-week change assessed after each MBCT session (up to 8 weeks) or weekly during wait-list (up to 8 weeks)
  Measured with the brooding subscale of the Ruminative Response Scale (RRS). The brooding subscale consists of 5 items. Scores range from 5-20. Higher scores indicate a higher level of depressive rumination.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Pro Persona, Nijmegen, Gelderland
  - Radboud University Medical Centre, Nijmegen, Gelderland

IPD SHARING:
Plan to Share IPD: Yes
The authors intend to make the data available to other researchers after completion of the study and will comply with open access procedures, including open access publishing, as much as possible.
Supporting Information: SAP, Analytic Code
Time Frame: The final report of the primary endpoint (assesment of whether MBCT-induced change in depressive symptoms is mediated by change in RNT) is expected December 2023.
Access Criteria: Restricted access. Meaning that interested researchers are welcome to contact us (authors) or the data-manager of the radboud data repository with requests for data. A team consisting of a data-manager and researchers will review the quality of the request and grant permission of the request is in accordance with the terms of use drafted by the Radboudumc and Radboud University.
URL: https://www.lcrdm.nl/

REFERENCES:
- [Derived] Lubbers J, Geurts DEM, Spinhoven P, Cladder-Micus MB, Ennen D, Speckens AEM, Spijker J. Rumination and Self-Compassion Moderate Mindfulness-Based Cognitive Therapy for Patients With Recurrent and Persistent Major Depressive Disorder: A Controlled Trial. Depress Anxiety. 2024 Nov 25;2024:3511703. doi: 10.1155/da/3511703. eCollection 2024. PMID 40226644

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT05802966/SAP_000.pdf